CLINICAL TRIAL: NCT02836184
Title: The Efficacy and Safety of Nicotinic Acid in the Hemodialysis Patients With Hyperphosphatemia
Brief Title: Nicotinic Acid in Hemodialysis Patients With Hyperphosphatemia
Acronym: NAHPH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiujiang No.1 People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaoran Feng, deputy director of nephrology division, Jiujiang No.1 People's Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016075
Record Dates: First submitted 2016-07-14; First posted 2016-07-18 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-07

CONDITIONS: Hyperphosphatemia
Keywords: Hemodialysis,Hyperphosphatemia,Nicotinic Acids
MeSH Terms: conditions — Hyperphosphatemia | interventions — Nicotinic Acids; Niacin; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (Active Comparator): Group treated with calcium carbonate for 6 weeks first,then switch to nicotinic acids treatment after 2 week of wash-out.
  Interventions: Drug: Calcium Carbonate
- nicotinic acids group (Experimental): Group treated with nicotinic acids for 6 weeks first,then switch to calcium carbonate treatment after 2 week of wash-out.
  Interventions: Drug: Nicotinic Acids

INTERVENTIONS:
Drug: Nicotinic Acids — Nicotinic acids is administered at an initial dosage of 50mg four times daily in the first week. If no significant side effects detected, the dosage will be titrated to 100mg five times daily within the second week and last to the end of study.
  Other Names: Niacin
  Arms: nicotinic acids group
Drug: Calcium Carbonate — Calcium Carbonate 500mg per oral, twice a day
  Other Names: Calcite
  Arms: control group

SUMMARY:
With calcium carbonate as the positive control drug, to observe the effectiveness and safety of nicotinic acid in hemodialysis patients with hyperphosphatemia

DETAILED DESCRIPTION:
Hyperphosphatemia is an important risk factor affecting long-term survival in patients with hemodialysis. Nicotinic acids, as well as its metabolites nicotinamide, were found to inhibit the sodium-phosphorus co-transporter on animal intestines. Several studies from other countries demonstrated that nicotinamide can reduce blood phosphorus levels in end-stage kidney disease patients. The purpose of this study was to investigate the effectiveness and safety of nicotinic acids on hyperphosphatemia in hemodialysis patients of ethnic Han live in China. The study is a prospective, randomized, double-blind, placebo-controlled crossover study. Eligible patients will be randomized to 6 wk of nicotinic acids or calcium carbonate. After a 2-wk washout period, patients switched to 6 wk of the alternative therapy. The primary measurement is the change in serum phosphorus during the whole term of each arm. Statistical analysis will be performed using two-sample paired-group t test.The significance level of the analysis was set to 0.05. All other adverse reactions will be analysed and reported, if there.

ELIGIBILITY:
Inclusion Criteria:

ethnic Han live in China, End-stage renal disease（ESRD）patients treated with hemodialysis ≥ 3 months, between 18 and 80 years of age, serum phosphorus > 1.78 mmol/L, capable of giving informed consent

Exclusion Criteria:

Be allergic to nicotinic acids, dysphagia, pregnant, current medication regimen including niacin or niacinamide active liver disease, peptic ulcer disease, full resection of parathyroid, malignancy, quit hemodialysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2016-07; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
change in serum phosphorus | Immediately after wash-out period and after 6 weeks of therapy.

SECONDARY OUTCOMES:
change in serum calcium | Immediately after wash-out period and after 6 weeks of therapy.
change in serum calcium-phosphorus product | Immediately after wash-out period and after 6 weeks of therapy.
change in intact parathyroid hormone | Immediately after wash-out period and after 6 weeks of therapy.
change in alkaline phosphatase | Immediately after wash-out period and after 6 weeks of therapy.
change in platelet count | Immediately after wash-out period and after 6 weeks of therapy.
change in serum uric acid | Immediately after wash-out period and after 6 weeks of therapy.
change in serum glucose | Immediately after wash-out period and after 6 weeks of therapy.
change in total cholesterol | Immediately after wash-out period and after 6 weeks of therapy.
change in triglyceride | Immediately after wash-out period and after 6 weeks of therapy.
change in high density lipoprotein cholesterol | Immediately after wash-out period and after 6 weeks of therapy.
change in low density lipoprotein cholesterol | Immediately after wash-out period and after 6 weeks of therapy.
change in serum glutamic-pyruvic transaminase | Immediately after wash-out period and after 6 weeks of therapy.
change in glutamic oxalacetic transaminase | Immediately after wash-out period and after 6 weeks of therapy.
change in bilirubin | Immediately after wash-out period and after 6 weeks of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoran Feng, MD,PHD, Principal Investigator — Department of Nephrology, Jiujiang NO.1 People's Hospital
Locations (1):
- Jiujiang NO.1 People's Hospital, Jiujiang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No